CLINICAL TRIAL: NCT05750225
Title: Retrospective, Non-interventional, Comparative Clinical Investigation of the Safety and Performance of 690AD and 690ADY Monofocal Intraocular Lens Implantation
Brief Title: Clinical Investigation of the Safety and Performance of Model 690AD and Model 690ADY Monofocal Intraocular Lens Implantation
Status: Completed | Type: Observational
Sponsor: Medicontur Medical Engineering Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: M_690AD/690ADY_HU_2203
Record Dates: First submitted 2023-02-09; First posted 2023-03-01 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2023-05

CONDITIONS: Cataract; Pseudophakia; Intraocular Lens Complication; Intraocular Lens Opacification
MeSH Terms: conditions — Cataract; Pseudophakia | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 690AD IOL: 50 eyes /patients implanted with 690AD IOL
  Interventions: Other: Standard of care; Other: Patient satisfaction questionnare
- 690ADY IOL: 50 eyes /patients implanted with 690ADY IOL
  Interventions: Other: Standard of care; Other: Patient satisfaction questionnare

INTERVENTIONS:
Other: Standard of care — 12 months after the IOL implantation: measurement of intraocular pressure, slitlamp and fundus examination, visual acuity, manifest refraction.
Other: Patient satisfaction questionnare — VFQ- 25 (Visual Function Questionnare) to be completed during 12 month visit.

SUMMARY:
Medicontur hydrophilic posterior chamber monofocal intraocular lens (IOLs) are indicated to improve vision at far distance in adults with cataract and/or ametropia (hyperopia, myopia), secondarily to removal of the crystalline lens.

The intraocular lens is intended to be surgically implanted into the eye with the purpose of restoring optical function in the aphakic eye to provide an optical system with high predictability of the precalculated dioptric power.

The study will be performed partially as a retrospective study with patients enrolled who had been implanted with 690AD or 690ADY IOLs mono- or binocularly between September 2021 - March 2022.

Data from five visits will be collected:

* Baseline preoperative (maximum 90 days prior to surgery)- retrospective
* IOL implantation Day 0 - retrospective
* Postoperative visit at Day 1 (+/- 0 days) - retrospective
* Postoperative visit at 1 month (+/- 2 weeks) - retrospective
* Postoperative visit at 12 months (+/- 3 months) - consent and prospective visit

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females above 18 years of age;
* Pseudophakic patients implanted with 690AD or 690ADY monofocal IOLs (implanted between September 2021 - March 2022);
* Diagnosis of cataract and/or ametropia (hyperopia, myopia);
* Subject who has signed an informed consent form.
* Patients who have participated in all visits that are subject to retrospective data collection.

Exclusion Criteria:

* - Patients who are not targeted to emmetropia.
* Patients with the following condition(s) at the time of the baseline visit:

  * Corneal astigmatism > 1.0 diopter
  * Uncontrolled diabetic retinopathy
  * Iris neovascularization
  * Congenital eye abnormality
  * Uncontrolled glaucoma
  * Pseudoexfoliation syndrome
  * Amblyopia
  * Uveitis
  * AMD (advanced AMD)
  * Retinal detachment
  * Prior ocular surgery in personal medical history
  * Previous laser treatment
  * Corneal diseases
  * Severe retinal diseases (dystrophy, degeneration)
  * High myopia
  * Inadequate visualization of the fundus on preoperative examination
  * Patients deemed by the clinical investigator because of any systemic disease
  * Pregnancy
  * Eye trauma in medical history
  * Current use of systemic steroids or topical ocular medication
* Patients with any eye condition that could affect vision in the opinion of the investigator at the time of the 12-month follow-up: (corneal ectasia, retinal diseases, glaucoma, uveitis, dry eye or amblyopia, etc.);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (18 years old and older) with cataract and/or ametropia (hyperopia, myopia), who have undergone monocular or binocular 690AD or 690ADY IOL implantation.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
CDVA | 12 months postoperatively
  Monocular corrected distance visual acuity (CDVA) To compare monocular corrected distance visual acuity (CDVA) between groups implanted with 690AD and 690ADY monofocal IOLs at 12 months postoperatively.

SECONDARY OUTCOMES:
UDVA | 12 months postoperatively
  Monocular uncorrected distance visual acuity (UDVA) To compare monocular uncorrected distance visual acuity (UDVA) between groups implanted with 690AD and 690ADY monofocal IOLs 12 months postoperatively.
UDVA and CDVA | 12 months postoperatively
  To compare percentage of eyes that achieve monocular UDVA and monocular CDVA within logMAR 0.0 or 0.3 between groups implanted with 690AD and 690ADY monofocal IOLs at 12 months postoperatively.
Spherical Equivalent | 12 months postoperatively
  Spherical Equivalent shall be used to calculate manifest residual refraction. To compare sphere, cylinder and axis of the eye between groups implanted with 690AD and 690ADY monofocal IOLs 12 months after IOL implantation.
Patient satisfaction | 12 months postoperatively
  Subjective perception of colour perception and scotopic vision shall be assessed by interviewing the patient using visual function questionnaire (VFQ-25 questionnaire) . To compare overall satisfaction, subjective perception of colour perception and scotopic vision between groups implanted with 690AD and 690ADY, postoperatively at 12 months.
Cylinder | 12 months postoperatively
  Cylinder shall be used to calculate manifest residual refraction.
Axis of the eye | 12 months postoperatively
  Axis of the eye shall be used to calculate manifest residual refraction.

OTHER OUTCOMES:
Intraoperative complications of cataract surgery | at Day1 postoperatively
  To verify that the frequency of the following complications does not exceed those stated in Acceptance criteria.
Postoperative complications of cataract surgery | at Month1 postoperatively
  To verify that the frequency of the following complications does not exceed those stated in Acceptance criteria.
Complications of IOL implantation | at Month12 postoperatively
  To verify that the frequency of the following complications does not exceed those stated in Acceptance criteria.

CONTACTS AND LOCATIONS:
Locations (2):
- Hungary (2):
  - Szabolcs-Szatmár-Bereg Megyei Kórházak és Egyetemi Oktatókórház, Jósa András Oktatókórház, Nyíregyháza
  - Pécsi Tudományegyetem, Klinikai Központ Szemészeti Klinika, Pécs